CLINICAL TRIAL: NCT05570526
Title: Effect Of Melatonin On The Clinical Outcome In Pediatric Hemodialysis Patients
Brief Title: Effect of Melatonin in Pediatric Hemodialysis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghadeer Amged, Demonstrator of clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RHDIRB2020110301 REC#99
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Hemodialysis Complication; Oxidative Stress; Inflammation
Keywords: Pediatric hemodialysis
MeSH Terms: conditions — Inflammation | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded, placebo-controlled trial.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group: (Experimental): 20 patients will receive oral melatonin 5mg tablets 1-hour before bedtime for 12 weeks.
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): 20 patients will receive one tablet of placebo 1-hour before bedtime for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Puritan's Pride ® Melatonin 5mg tablets orally once daily.
  Arms: Intervention group:
Other: Placebo — Placebo tablet once daily.
  Arms: Placebo

SUMMARY:
A Prospective, randomized, double-blinded, placebo-controlled trial will be conducted at the pediatric dialysis unit, Children's Hospital, Ain Shams University in order to investigate the benefits of melatonin supplementation on oxidative stress, inflammation and to assess sleep quality by using PSQI questionnaire in pediatric hemodialysis patients.

DETAILED DESCRIPTION:
1. Patients will be recruited and evaluated for eligibility.
2. Patients who meet the eligibility criteria will be randomly assigned to either placebo or intervention group.
3. Patient demographics, clinical characteristics and full medical and medication history: will be obtained at baseline and every 4 weeks after the beginning of the study.
4. Blood samples will be withdrawn from each patient before the dialysis session for assay of each of the following:

1.Oxidative stress marker malondialdehyde (MDA) by ELISA assay. 2. Inflammatory marker level nuclear factor kappa B (NF-KB) by ELISA assay 3. Complete blood picture (CBC). 4. Lipid profile (total cholesterol(TC), triglycerides(TG), high-density lipoprotein (HDL) and low-density lipoprotein (LDL) 5)Safety will be assessed weekly after the beginning of the study by monitoring the side effects or any adverse drug reactions.

* A total of (40) patients on regular HD will be enrolled in the study. These patients will be randomly assigned in a 1:1 ratio into two groups:

  * The first group (n=20):The patients in the first group will receive a total daily dose of 5mg of melatonin tablets 1-hour before bedtime for 12 weeks.
  * The second group (n=20): The patients will receive one tablet of placebo for the same duration.
* All subjects will sign an informed consent statement prior to inclusion in the study.
* All subjects will be followed up weekly for 12 weeks and blood samples will be withdrawn at baseline and the end of the study.

ELIGIBILITY:
All patients will be assessed for eligibility according to the following inclusion and exclusion criteria:

Inclusion Criteria:

1. Male or female patients age from 6-18 years old.
2. Undergoing regular HD for at least 6 months prior to enrollment
3. Not enrolled in any other clinical trial.
4. Judged by the physician to be physically stable

Exclusion Criteria:

1. Patients receiving anti-epileptics.
2. Patients with some autoimmune conditions as SLE, RA or post-organ transplant
3. Patients taking immunosuppressants.
4. Patients taking warfarin.
5. Patients receiving vitamin E, green tea or zinc during the past 3 months
6. Patients with malignancy and/or active inflammatory disease
7. Patients with mal absorption, mental retardation or psychiatric illness.
8. Patients who had hemorrhagic episodes or received blood transfusion in the past 3 months prior to the enrollment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Malondialdehyde (MDA) level. | At baseline and at 12 weeks.
  Oxidative stress marker

SECONDARY OUTCOMES:
Change in baseline nuclear factor kappa B (NF-KB) level. | At baseline and at 12 weeks.
  Inflammatory marker
Change in sleep quality by using Pittsburgh Sleep Quality Index (PSQI) questionnaire | At baseline and at 12 weeks.
  Sleep quality assessment using the validated Arabic version of PSQI questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasseya, Egypt

REFERENCES:
- [Derived] Sayed GA, El Borolossy RM, Said RM, Shaheen SM. Evaluating the antioxidant and anti-inflammatory effect of melatonin in pediatric hemodialysis patients: a randomized, placebo-controlled trial. Sci Rep. 2026 Jan 21. doi: 10.1038/s41598-025-34264-0. Online ahead of print. PMID 41565787